CLINICAL TRIAL: NCT01093703
Title: Randomized Trial to Explore the Effect of Chronotherapy Versus Conventional BP Control to Correct Abnormal Circadian BP Pattern and Improve Allograft Function in Kidney Transplant Recipients
Brief Title: Chronotherapy Versus Conventional BP Control to Correct Abnormal Circadian BP Pattern in Kidney Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Hani M. Wadei, Cons-Nephrology, Mayo Clinic
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 08-005049
Record Dates: First submitted 2010-03-24; First posted 2010-03-26 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Blood Pressure Control; Kidney Transplant Recipient
Keywords: kidney transplantation; hypertension; chronotherapy; graft function; circadian pattern
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional Therapy (No Intervention): In the conventional therapy group, no medication changes other than the ones needed to achieve target awake average SBP will be undertaken. Time at which patients are taking their BP medications will be recorded.
- Intensive Therapy (Active Comparator): In the intensive therapy group, BP medications will be adjusted to both control awake average systolic BP to target and to cover the overnight period in an attempt to control nocturnal hypertension.
  Interventions: Other: Medication Adjustment

INTERVENTIONS:
Other: Medication Adjustment — 1. Awake SBP≤135/85mmHg and patient is on once daily medications: Switch BP medications to pm period.
  2. Awake SBP SBP≤135/85mmHg and patient is on bid medications (e.g. metoprolol bid): Increase pm dose of the medication. If medication is already is at maximal dose or there is contraindication for increasing the dose (e.g. bradycardia), add another BP medicine in the evening time.
  3. Awake SBP≤135/85mmHg and patient is not on anti-hypertensive medications: Add BP medication at the pm period.
  4. Awake SBP>135/85mmHg: increase dose of antihypertensive medications or add more medications. All medications to be given in the evening time.
  Arms: Intensive Therapy

SUMMARY:
The purpose of this study is to identify and manage factors related to blood pressure control that impact organ function and survival in kidney transplant recipients. Loss of the circadian (relating to a 24-hour rhythm) blood pressure pattern is common in kidney transplant recipients and is associated with poor allograft kidney function. It is still unclear if restoring the normal day-night blood pressure (BP) pattern will translate into better allograft outcome. Although studies in patients with and without chronic kidney disease indicate that restoration of the normal nocturnal (night) dipping in BP is possible by changing the timing of the BP medications to cover the overnight period (chronotherapy), this has not been tested in kidney transplant patients.

DETAILED DESCRIPTION:
The challenge in kidney transplantation is to identify and manage factors that impact allograft function and survival. Loss of the circadian blood pressure pattern is common in kidney transplant recipients and is associated with poor allograft kidney function. Nevertheless, it is unclear if restoring the normal day-night BP pattern will translate into better allograft outcome. Although studies in patients with and without chronic kidney disease indicate that restoration of the normal nocturnal dipping in BP is possible by changing the timing of the BP medications to cover the overnight period (chronotherapy), this has not been tested in kidney transplant patients. This exploratory study is driven by the hypothesis that chronotherapy will restore the normal circadian BP pattern and will translate into better allograft function and into lower LVM 1-year from transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Recipient of a kidney transplant.
* Age≥18 years.
* Stable allograft function.
* Ability to give informed consent.

Exclusion Criteria:

* Multiorgan transplant recipients.
* Kidney transplant recipients with poor allograft function.
* Documented history of obstructive sleep apnea.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2008-12; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Percent drop in mean SBP at night-time compared to mean SBP in day-time | 1 year
Glomerular filtration rate | 1 year

SECONDARY OUTCOMES:
Awake mean SBP | 1 year
Presence of abnormal circadian BP pattern in recipients on steroid free and CIN free IS | 1 year
Change in LVM | 1 year
Urinary microalbumin excretion | 4 months & 1 year
Long term renal function | 2 years
Cardiovascular events (stroke, heart failure, myocardial infarction) | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States

REFERENCES:
- [Background] Mange KC, Cizman B, Joffe M, Feldman HI. Arterial hypertension and renal allograft survival. JAMA. 2000 Feb 2;283(5):633-8. doi: 10.1001/jama.283.5.633. PMID 10665703
- [Background] Kasiske BL, Anjum S, Shah R, Skogen J, Kandaswamy C, Danielson B, O'Shaughnessy EA, Dahl DC, Silkensen JR, Sahadevan M, Snyder JJ. Hypertension after kidney transplantation. Am J Kidney Dis. 2004 Jun;43(6):1071-81. doi: 10.1053/j.ajkd.2004.03.013. PMID 15168388
- [Background] Opelz G, Dohler B; Collaborative Transplant Study. Improved long-term outcomes after renal transplantation associated with blood pressure control. Am J Transplant. 2005 Nov;5(11):2725-31. doi: 10.1111/j.1600-6143.2005.01093.x. PMID 16212633
- [Background] Clement DL, De Buyzere ML, De Bacquer DA, de Leeuw PW, Duprez DA, Fagard RH, Gheeraert PJ, Missault LH, Braun JJ, Six RO, Van Der Niepen P, O'Brien E; Office versus Ambulatory Pressure Study Investigators. Prognostic value of ambulatory blood-pressure recordings in patients with treated hypertension. N Engl J Med. 2003 Jun 12;348(24):2407-15. doi: 10.1056/NEJMoa022273. PMID 12802026
- [Background] Shimada K, Kawamoto A, Matsubayashi K, Nishinaga M, Kimura S, Ozawa T. Diurnal blood pressure variations and silent cerebrovascular damage in elderly patients with hypertension. J Hypertens. 1992 Aug;10(8):875-8. PMID 1325522
- [Background] Verdecchia P, Porcellati C, Schillaci G, Borgioni C, Ciucci A, Battistelli M, Guerrieri M, Gatteschi C, Zampi I, Santucci A, Santucci C, Reboldi G, et al. Ambulatory blood pressure. An independent predictor of prognosis in essential hypertension. Hypertension. 1994 Dec;24(6):793-801. doi: 10.1161/01.hyp.24.6.793. PMID 7995639
- [Background] Haydar AA, Covic A, Jayawardene S, Agharazii M, Smith E, Gordon I, O'Sullivan H, Goldsmith DJ. Insights from ambulatory blood pressure monitoring: diagnosis of hypertension and diurnal blood pressure in renal transplant recipients. Transplantation. 2004 Mar 27;77(6):849-53. doi: 10.1097/01.tp.0000115345.16853.51. PMID 15077025
- [Background] Agarwal R, Andersen MJ. Prognostic importance of ambulatory blood pressure recordings in patients with chronic kidney disease. Kidney Int. 2006 Apr;69(7):1175-80. doi: 10.1038/sj.ki.5000247. PMID 16467785
- [Background] Lurbe E, Redon J, Kesani A, Pascual JM, Tacons J, Alvarez V, Batlle D. Increase in nocturnal blood pressure and progression to microalbuminuria in type 1 diabetes. N Engl J Med. 2002 Sep 12;347(11):797-805. doi: 10.1056/NEJMoa013410. PMID 12226150
- [Background] Davidson MB, Hix JK, Vidt DG, Brotman DJ. Association of impaired diurnal blood pressure variation with a subsequent decline in glomerular filtration rate. Arch Intern Med. 2006 Apr 24;166(8):846-52. doi: 10.1001/archinte.166.8.846. PMID 16636209
- [Background] Kapa S, Sert Kuniyoshi FH, Somers VK. Sleep apnea and hypertension: interactions and implications for management. Hypertension. 2008 Mar;51(3):605-8. doi: 10.1161/HYPERTENSIONAHA.106.076190. Epub 2008 Jan 28. No abstract available. PMID 18227409
- [Background] Pennestri MH, Montplaisir J, Colombo R, Lavigne G, Lanfranchi PA. Nocturnal blood pressure changes in patients with restless legs syndrome. Neurology. 2007 Apr 10;68(15):1213-8. doi: 10.1212/01.wnl.0000259036.89411.52. PMID 17420405
- [Background] Khot UN, Binkley PF, Haas GJ, Starling RC. Prospective study of the circadian pattern of blood pressure after heart transplantation. J Heart Lung Transplant. 1996 Apr;15(4):350-9. PMID 8732593
- [Background] Taler SJ, Textor SC, Canzanello VJ, Wilson DJ, Wiesner RH, Krom RA. Loss of nocturnal blood pressure fall after liver transplantation during immunosuppressive therapy. Am J Hypertens. 1995 Jun;8(6):598-605. doi: 10.1016/0895-7061(95)00077-3. PMID 7544983
- [Background] Toprak A, Koc M, Tezcan H, Ozener IC, Oktay A, Akoglu E. Night-time blood pressure load is associated with higher left ventricular mass index in renal transplant recipients. J Hum Hypertens. 2003 Apr;17(4):239-44. doi: 10.1038/sj.jhh.1001536. PMID 12692568
- [Background] Wadei HM, Amer H, Taler SJ, Cosio FG, Griffin MD, Grande JP, Larson TS, Schwab TR, Stegall MD, Textor SC. Diurnal blood pressure changes one year after kidney transplantation: relationship to allograft function, histology, and resistive index. J Am Soc Nephrol. 2007 May;18(5):1607-15. doi: 10.1681/ASN.2006111289. Epub 2007 Apr 4. PMID 17409307
- [Background] Covic A, Gusbeth-Tatomir P, Mardare N, Buhaescu I, Goldsmith DJ. Dynamics of the circadian blood pressure profiles after renal transplantation. Transplantation. 2005 Nov 15;80(9):1168-73. doi: 10.1097/01.tp.0000167003.97452.a8. PMID 16314781
- [Background] Logan AG, Tkacova R, Perlikowski SM, Leung RS, Tisler A, Floras JS, Bradley TD. Refractory hypertension and sleep apnoea: effect of CPAP on blood pressure and baroreflex. Eur Respir J. 2003 Feb;21(2):241-7. doi: 10.1183/09031936.03.00035402. PMID 12608436
- [Background] Minutolo R, Gabbai FB, Borrelli S, Scigliano R, Trucillo P, Baldanza D, Laurino S, Mascia S, Conte G, De Nicola L. Changing the timing of antihypertensive therapy to reduce nocturnal blood pressure in CKD: an 8-week uncontrolled trial. Am J Kidney Dis. 2007 Dec;50(6):908-17. doi: 10.1053/j.ajkd.2007.07.020. PMID 18037091
- [Background] Hermida RC, Ayala DE, Fernandez JR, Calvo C. Chronotherapy improves blood pressure control and reverts the nondipper pattern in patients with resistant hypertension. Hypertension. 2008 Jan;51(1):69-76. doi: 10.1161/HYPERTENSIONAHA.107.096933. Epub 2007 Oct 29. PMID 17968001
- [Background] Hermida RC, Ayala DE, Calvo C, Lopez JE, Mojon A, Fontao MJ, Soler R, Fernandez JR. Effects of time of day of treatment on ambulatory blood pressure pattern of patients with resistant hypertension. Hypertension. 2005 Oct;46(4):1053-9. doi: 10.1161/01.HYP.0000172757.96281.bf. Epub 2005 Aug 8. PMID 16087787
- [Background] Hermida RC, Ayala DE, Calvo C. Administration-time-dependent effects of antihypertensive treatment on the circadian pattern of blood pressure. Curr Opin Nephrol Hypertens. 2005 Sep;14(5):453-9. doi: 10.1097/01.mnh.0000174144.07174.74. PMID 16046904
- [Background] Hermida RC, Calvo C, Ayala DE, Lopez JE. Decrease in urinary albumin excretion associated with the normalization of nocturnal blood pressure in hypertensive subjects. Hypertension. 2005 Oct;46(4):960-8. doi: 10.1161/01.HYP.0000174616.36290.fa. Epub 2005 Sep 6. PMID 16144987
- [Background] Gali B, Whalen FX Jr, Gay PC, Olson EJ, Schroeder DR, Plevak DJ, Morgenthaler TI. Management plan to reduce risks in perioperative care of patients with presumed obstructive sleep apnea syndrome. J Clin Sleep Med. 2007 Oct 15;3(6):582-8. PMID 17993039
- See also: Related Info — http://www.mayoclinic.org/